CLINICAL TRIAL: NCT01618565
Title: Objective Structured Assessment of Technical Skills (OSATS) Evaluation of Theoretical Versus Hands-On Training of Shoulder Dystocia Management: a Randomized Trial
Brief Title: Objective Structured Assessment of Technical Skills (OSATS) Evaluation of Shoulder Dystocia Management
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clemens Tempfer (Other)
Responsible Party: Sponsor-Investigator, Clemens Tempfer, Department head ObGyn, Ruhr University of Bochum
Organization: Ruhr University of Bochum (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SD-1
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Shoulder Dystocia
Keywords: shoulder dystocia; training; To assess the effectiveness of hands-on training versus expert demonstration
MeSH Terms: conditions — Shoulder Dystocia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hands-On Training (Experimental): 30 minutes hands-on training of maneuvers to manage shoulder dystocia
  Interventions: Procedure: Hands-On Training
- Demonstration (Active Comparator): 30 minutes passive training by watching an expert instructor explain and perform maneuvers to manage shoulder dystocia
  Interventions: Procedure: Demonstration

INTERVENTIONS:
Procedure: Hands-On Training — one-time, 30 minute hands-on training
  Arms: Hands-On Training
Procedure: Demonstration — 30 minutes passive training
  Arms: Demonstration

SUMMARY:
This trial tests whether hands-on training is superior to expert demonstration regarding the management of shoulder dystocia (stuck shoulder) during delivery on a training model.

DETAILED DESCRIPTION:
We prospectively randomize probands to a 30 min hands-on (group 1) and a 30 min demonstration (group 2) training session teaching a standardized SD algorithm scheme on a pelvic training model. Probands are tested with a 22 item Objective Structured Assessment of Technical Skills (OSATS) scoring system after training and 72 hours thereafter. OSATS scores are the primary outcome. Performance time (PT), self assessment (SA), confidence (CON), and global rating scale (GRS) are the secondary outcomes. Statistics will beperformed using Mann-Whitney U-test, chi-square test, and multivariable logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
OSATS Score | 30 minutes
  Probands are tested with a 22 item Objective Structured Assessment of Technical Skills (OSATS) scoring system after training and 72 hours thereafter.

SECONDARY OUTCOMES:
Performance Time | 30 minutes
  Time probands need to perform all test tasks
Global Rating Scale | 30 minutes
  Predefined score including confidence, speed, and manual capacity to perform test tasks

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Dept. OBGYN Ruhr University Bochum, Herne
  - Dept. OBGYN, Ruhr University Bochum, Herne

REFERENCES:
- [Result] Buerkle B, Pueth J, Hefler LA, Tempfer-Bentz EK, Tempfer CB. Objective structured assessment of technical skills evaluation of theoretical compared with hands-on training of shoulder dystocia management: a randomized controlled trial. Obstet Gynecol. 2012 Oct;120(4):809-14. doi: 10.1097/AOG.0b013e31826af9a9. PMID 22996098